CLINICAL TRIAL: NCT00630721
Title: Characterization of Interferon Beta -1b-Induced Tolerizing Effect in Dendritic Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 07-0941
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IFNbeta-1b (Other): no drug was given under study. patients already taking IFNbeta-1b were enrolled for blood draw only.
  Interventions: Other: IFNbeta-1b

INTERVENTIONS:
Other: IFNbeta-1b — no drug was given under study arm. only blood draw on patients already on IFNbeta-1b.

SUMMARY:
Determine the in-vivo mechanism of action of INF-B-1b as it's mechanisms of action are not completely understood. We propose that high dose exogenous recombinant IFN-B-1b induces tolerizing effect on DC-dependent T-cell differentiation in patients with MS by inducing the expression of SOCS3 in DCs.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MS
* Age 18-60 years, inclusive
* Expanded disability status of 0-6.5
* Give written informed consent prior to any testing under this protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2007-09; Primary Completion 2010-05-15 (Actual); Study Completion 2011-03-15 (Actual)

PRIMARY OUTCOMES:
Determine the effect of IFN-B-1b-induced SOCS3 upregulation in DCs' on their maturation and the capacity to present | 2 years

SECONDARY OUTCOMES:
Characterize the effect of IFN-1b-induced SOCS3 expression in DCs on Th1/Th2 cell differentiation and T-cell cytokine transcription. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Silva Markovic-Plese, MD, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States